CLINICAL TRIAL: NCT03740997
Title: A Phase 4, Open-Label, Non-Randomized, Multicenter Study to Evaluate Safety and Efficacy of Intravenous Administration of OPTISON™ for Contrast- Enhanced Echocardiography in Pediatric Patients
Brief Title: Study to Determine Safety and Dosage of OPTISON in Pediatric Participants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Laboratory Corporation of America (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GE-191-008
Record Dates: First submitted 2018-10-31; First posted 2018-11-14 (Actual); Results first posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-03

CONDITIONS: Transthoracic Echocardiography; Suspected or Known Structural or Functional Cardiac Abnormality
Keywords: Contrast-enhanced echocardiography (CE-ECHO); Transthoracic echocardiogram; Child; Left ventricular opacification (LVO); Left ventricular ejection fraction (LVEF); Left ventricular endocardial border delineation (LV EBD)
MeSH Terms: interventions — FS 069

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Body Weight Group <=40 kg: OPTISON (Experimental): Participants with body weight greater than or equal to (>=) 20 to less than or equal to (<=) 28 kilograms (kg) received OPTISON 0.1 milliliter (mL; dose level 1) or 0.2 mL (dose level 2); and participants with body weight greater than (>) 28 to <=40 kg received OPTISON 0.2 mL (dose level 1) or 0.3 mL (dose level 2) intravenous (IV) injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose for body weight >=20 to <=28 kg and >28 to <=40 kg was 1.0 mL and 1.5 mL per dose level, respectively.
  The treated subjects received both dose levels. Per protocol, up to 3 injections per dose level were allowed for acquiring different imaging views. A maximum of 2 injections was recorded in the treated population.
  Interventions: Drug: Optison
- Body Weight Group >40 kg: OPTISON (Experimental): Participants with body weight >40 kg received OPTISON 0.2 (dose level 1) or 0.4 mL (dose level 2) IV injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose was 1.8 mL per dose level.
  The treated subjects received both dose levels. Per protocol, up to 3 injections per dose level were allowed for acquiring different imaging views. A maximum of 2 injections was recorded in the treated population.
  Interventions: Drug: Optison

INTERVENTIONS:
Drug: Optison — Optison is administered intravenously
  Other Names: Perflutren Microspheres Injectable Suspension, USP

SUMMARY:
Study to determine the safety and appropriate dosage of OPTISON in pediatric participants since OPTISON has been tested in adult participants only during the clinical development

ELIGIBILITY:
Inclusion Criteria:

* The participant was between ≥9 and <18 years of age and weighs ≥20 kg.
* The participant was clinically indicated to undergo a transthoracic echocardiogram.
* The participant had a suboptimal non-contrast echocardiogram defined as ≥2 contiguous segments in any given view that cannot be visualized.
* The participant was able to comply with study procedures.
* A parent or legal guardian of the participant had signed and dated an informed consent form.
* Post-menarchal female participants must have had a negative urine pregnancy test at screening and at pre-dose on the day of OPTISON administration.
* Post-menarchal female participants must have been practicing abstinence, or be using an effective form of birth control (e.g., intrauterine device, oral contraceptives, contraceptive implants or injections, diaphragm with spermicide, cervical cap, or consort use of condom) for at least 30 days before being enrolled in the study

Exclusion Criteria:

* The participant was previously enrolled in this study.
* The participant received an investigational medicinal product within 30 days before or is scheduled to receive one from time of entry into this study until completion of the follow-up period proposed for this study.
* The participant had a known or suspected hypersensitivity to any of the components of OPTISON, blood, blood products, or albumin.
* The participant had pulmonary hypertension or unstable cardiopulmonary conditions.
* The participant had severe liver disease based on medical history.
* The participant had a recent (<6 months) neurological event.
* The participant presented any clinically active, serious, life-threatening disease, with a life expectancy of less than 1 month or where study participation may compromise the management of the participant or other reason that in the judgment of the investigator makes the participant unsuitable for participation in the study.
* The participant was a pregnant or lactating female, or was a female of childbearing potential not using an acceptable form of birth control (negative urine pregnancy test was also required).

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Thompson, MD, PhD, Study Director — GE Healthcare
Locations (8):
- United States (8):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - MCG Health, Inc., Augusta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Cohen Children's Medical Center of New York, Lake Success, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Baylor College of Medicine, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted between 01 December 2020 to 30 March 2023 at 8 centers in the United States.
Pre-assignment Details: A total 39 participants were enrolled into the study, of which 37 received OPTISON injections according to body weight (less than or equal to [<=40] kilograms [kg] [included participants with body weight more than or equal to [>=] 20 to <=28 kg and greater than [>] 28 to <=40 kg] and >40 kg). As pre planned in Statistical Analysis Plan, data were collected, analyzed and presented for two body weight categories (<= 40 kg and >40 kg) only in all sections of the result.
Groups:
- Body Weight Group >40 kg: OPTISON: Participants with body weight >40 kg received OPTISON 0.2 (dose level 1) or 0.4 mL (dose level 2) IV injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose was 1.8 mL per dose level.
  The 37 treated subjects received both dose levels. Per protocol, up to 3 injections per dose level were allowed for acquiring different imaging views. A maximum of 2 injections was recorded in the treated population.
- Body Weight Group <=40 kg: OPTISON: Participants with body weight >=20 to <=28 kg received OPTISON 0.1 milliliter (mL; dose level 1) or 0.2 mL (dose level 2); and participants with body weight >28 to <=40 kg received OPTISON 0.2 mL (dose level 1) or 0.3 mL (dose level 2) intravenous (IV) injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose for body weight >=20 to <=28 kg and >28 to <=40 kg was 1.0 mL and 1.5 mL per dose level, respectively.
  The 37 treated subjects received both dose levels. Per protocol, up to 3 injections per dose level were allowed for acquiring different imaging views. A maximum of 2 injections was recorded in the treated population.
Period: Overall Study
Arm/Group | Body Weight Group >40 kg: OPTISON | Body Weight Group <=40 kg: OPTISON
Started | 31 | 8
Safety Population (Treated) (The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study.) | 29 | 8
Per-protocol (PP) Population (The PP population consisted of all participants who had available non-contrast harmonic images and OPTISON-enhanced echocardiographic images, irrespective of the quality of contrast-enhanced (CE)-echo and who did not have an important protocol deviation impacting the study primary endpoint.) | 23 | 7
Completed | 29 | 8
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Participant was unable to complete study procedures | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study.
Groups:
- Body Weight Group <=40 kg: OPTISON: Participants with body weight >=20 to <=28 kg received OPTISON 0.1 mL (dose level 1) or 0.2 mL (dose level 2); and participants with body weight >28 to <=40 kg received OPTISON 0.2 mL (dose level 1) or 0.3 mL (dose level 2) IV injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose for body weight >=20 to <=28 kg and >28 to <=40 kg was 1.0 mL and 1.5 mL per dose level, respectively.
- Body Weight Group >40 kg: OPTISON: Participants with body weight >40 kg received OPTISON 0.2 (dose level 1) or 0.4 mL (dose level 2) IV injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose was 1.8 mL per dose level.
- Total: Total of all reporting groups
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON | Total
Number analyzed (Participants) | 8 | 29 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (1.60) | 14.3 (2.09) | 13.4 (2.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 11 | 14
  Male | 5 | 18 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 15 | 18
  Not Hispanic or Latino | 5 | 13 | 18
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 6 | 20 | 26
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Total Visualization Score of Qualitative Endocardial Border Delineation (EBD) of the 12 Segments of the Left Ventricle (LV) Wall in Standard Apical 4-chamber (A4C) and Apical 2-chamber (A2C)
Description: Visualization of each of the 12 segments of the LV wall in standard A4C and A2C views were measured by the qualitative EBD visualization scale: score 0 =no visualization of the LV endocardial border; 1 =poor visualization; 2 =fair visualization; 3 =good/optimal visualization. The total LV EBD score was calculated as the sum of the individual scores assigned to each of the 12 LV wall segment and the total score ranged from 0 (no visualization of the LV endocardial border) to 36 (good/optimal visualization). A higher score indicated better visualization. The total score of qualitative EBD visualization scale were reported by reader (independent blinded), non-contrast and dose levels.
Time Frame: Images were captured during the study echocardiogram (0 to 30 minutes) on Day 1 and blinded image evaluations (BIE) were carried out at the study core laboratory following image transfer
Population: PP population consisted of all participants who had available non-contrast harmonic images and OPTISON-enhanced echocardiographic images, irrespective of the quality of CE-echo and who did not have an important protocol deviation impacting study primary endpoint. Each participant underwent an echocardiographic procedure first without contrast administration, then intravenous bolus injection of OPTISON. Here, "Number Analyzed" signifies participants who were evaluable for specified categories.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 7 | 23
score on a scale
  Reader 1: Non-contrast | 15.9 (5.73) | 10.0 (7.02)
  Reader 1: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 1: OPTISON Dose Level 1 | 31.3 (6.53) | 26.6 (12.50)
  Reader 1: OPTISON Dose Level 2 | 35.1 (2.27) | 28.6 (10.36)
  Reader 2: Non-contrast | 13.4 (2.57) | 8.5 (6.49)
  Reader 2: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 2: OPTISON Dose Level 1 | 32.8 (1.47) | 28.1 (10.34)
  Reader 2: OPTISON Dose Level 2 | 35.4 (0.79) | 29.7 (10.10)
  Reader 3: Non-contrast | 21.3 (7.13) | 12.5 (9.56)
  Reader 3: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 3: OPTISON Dose Level 1 | 32.5 (3.73) | 27.8 (10.40)
  Reader 3: OPTISON Dose Level 2 | 33.4 (2.07) | 28.3 (8.41)
Statistical Analysis 1: Comparison: Body Weight Group <=40 kg: OPTISON; Reader 1: Difference Between Non-contrast and OPTISON Dose Level 1; Test type: Other; p = 0.0008, Paired t-test; Mean Difference (Net) = 16.2, 95% CI 2-sided [10.44 to 21.89], Standard Deviation 5.46
Statistical Analysis 2: Comparison: Body Weight Group >40 kg: OPTISON; Reader 1: Difference Between Non-contrast and OPTISON Dose Level 1; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 17.1, 95% CI 2-sided [11.11 to 23.07], Standard Deviation 13.49
Statistical Analysis 3: Comparison: Body Weight Group <=40 kg: OPTISON; Reader 1: Difference Between Non-contrast and OPTISON Dose Level 2; Test type: Other; p = 0.0002, Paired t-test; Mean Difference (Net) = 19.3, 95% CI 2-sided [13.28 to 25.30], Standard Deviation 6.50
Statistical Analysis 4: Comparison: Body Weight Group >40 kg: OPTISON; Reader 1: Difference Between Non-contrast and OPTISON Dose Level 2; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 18.5, 95% CI 2-sided [13.47 to 23.57], Standard Deviation 11.68
Statistical Analysis 5: Comparison: Body Weight Group <=40 kg: OPTISON; Reader 2: Difference Between Non-contrast and OPTISON Dose Level 1; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 19.8, 95% CI 2-sided [16.62 to 23.05], Standard Deviation 3.06
Statistical Analysis 6: Comparison: Body Weight Group >40 kg: OPTISON; Reader 2: Difference Between Non-contrast and OPTISON Dose Level 1; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 20.1, 95% CI 2-sided [14.16 to 26.03], Standard Deviation 13.38
Statistical Analysis 7: Comparison: Body Weight Group <=40 kg: OPTISON; Reader 2: Difference Between Non-contrast and OPTISON Dose Level 2; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 22.0, 95% CI 2-sided [19.44 to 24.56], Standard Deviation 2.77
Statistical Analysis 8: Comparison: Body Weight Group >40 kg: OPTISON; Reader 2: Difference Between Non-contrast and OPTISON Dose Level 2; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 21.2, 95% CI 2-sided [15.45 to 26.99], Standard Deviation 13.34
Statistical Analysis 9: Comparison: Body Weight Group <=40 kg: OPTISON; Reader 3: Difference Between Non-contrast and OPTISON Dose Level 1; Test type: Other; p = 0.0268, Paired t-test; Mean Difference (Net) = 11.8, 95% CI 2-sided [2.02 to 21.64], Standard Deviation 9.35
Statistical Analysis 10: Comparison: Body Weight Group >40 kg: OPTISON; Reader 3: Difference Between Non-contrast and OPTISON Dose Level 1; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 16.1, 95% CI 2-sided [9.45 to 22.82], Standard Deviation 15.08
Statistical Analysis 11: Comparison: Body Weight Group <=40 kg: OPTISON; Reader 3: Difference Between Non-contrast and OPTISON Dose Level 2; Test type: Other; p = 0.0028, Paired t-test; Mean Difference (Net) = 12.1, 95% CI 2-sided [6.04 to 18.24], Standard Deviation 6.59
Statistical Analysis 12: Comparison: Body Weight Group >40 kg: OPTISON; Reader 3: Difference Between Non-contrast and OPTISON Dose Level 2; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Net) = 15.8, 95% CI 2-sided [10.04 to 21.61], Standard Deviation 13.37

2. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily had to have causal relationship with treatment. TEAEs were defined as AEs that starts or worsens at or after the time of first dosing of OPTISON.
Time Frame: 0- 72 hours
Population: The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
Participants | 4 | 9

3. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Systolic and diastolic blood pressure were measured from the arm contra-lateral to the site of OPTISON administration whenever possible and before measurement, participants rested for at least 5 minutes (if possible).
Time Frame: Baseline (pre-dose), and at 10 and 60 minutes post last dose on Day 1
Population: The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study. Here, "Number Analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
millimeter of mercury (mmHg)
  Systolic Blood Pressure: Change at 10 Minutes Post Last Dose | -3.3 (8.21) | -4.6 (10.46)
  Systolic Blood Pressure: Change at 60 Minutes Post Last Dose: number analyzed (Participants) | 8 | 28
  Systolic Blood Pressure: Change at 60 Minutes Post Last Dose | -4.8 (4.68) | -3.8 (12.01)
  Diastolic Blood Pressure: Change at 10 Minutes Post Last Dose | -2.8 (5.37) | -2.5 (11.67)
  Diastolic Blood Pressure: Change at 60 Minutes Post Last Dose: number analyzed (Participants) | 8 | 28
  Diastolic Blood Pressure: Change at 60 Minutes Post Last Dose | -1.8 (4.65) | -1.1 (9.95)

4. Secondary Outcome: Change From Baseline in Heart Rate
Description: Before heart rate was measured, participants rested for at least 5 minutes (if possible).
Time Frame: Baseline (pre-dose), and at 10 and 60 minutes post last dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
beats per minute
  Change at 10 Minutes Post Last Dose | -3.1 (7.90) | -4.9 (9.79)
  Change at 60 Minutes Post Last Dose: number analyzed (Participants) | 8 | 28
  Change at 60 Minutes Post Last Dose | -3.8 (15.69) | -2.1 (11.31)

5. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Before respiratory rate was measured, participants rested for at least 5 minutes (if possible).
Time Frame: Baseline (pre-dose), and at 10 and 60 minutes post last dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
breaths per minute
  Change at 10 Minutes Post Last Dose | -0.8 (3.99) | -0.2 (3.71)
  Change at 60 Minutes Post Last Dose: number analyzed (Participants) | 8 | 28
  Change at 60 Minutes Post Last Dose | -0.8 (1.49) | -1.5 (4.30)

6. Secondary Outcome: Change From Baseline in Oxygen Saturation as Measured by Pulse Oximetry
Description: Oxygen saturation was measured by pulse oximetry. Before oxygen saturation was measured, participants rested for at least 5 minutes (if possible).
Time Frame: Baseline (pre-dose), and at 10 and 60 minutes post last dose on Day 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of oxygen saturation
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
percentage of oxygen saturation
  Change at 10 Minutes Post Last Dose | 0.0 (1.20) | 0.1 (1.19)
  Change at 60 Minutes Post Last Dose: number analyzed (Participants) | 8 | 28
  Change at 60 Minutes Post Last Dose | -0.5 (2.07) | -0.2 (1.32)

7. Secondary Outcome: Number of Participants With Clinically Significant Abnormality in Physical Examination Findings
Description: Participants underwent assessments including general appearance, respiratory, cardiovascular and neurological (motor function, level of consciousness, sensory function) examination. Any abnormal clinically significant physical examination findings were based on investigator decision.
Time Frame: From first dose (Day 1) of study drug to 60 minutes post last dose on Day 1
Population: The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
Participants | 0 | 0

8. Secondary Outcome: Change From Baseline in 12-lead Electrocardiograms (ECGs) Parameters
Description: Change from baseline in PR, QRS, QT, Bazett's formula corrected QT (QTcB), Fridericia's formula corrected QT (QTcF) and RR intervals expressed in millisecond (ms) were reported.
Time Frame: Baseline (pre-dose), and at 10 and 30 minutes post last dose on Day 1
Population: The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 8 | 29
milliseconds (ms)
  PR Interval: Change at 10 Minutes Post Last Dose | -2.5 (4.14) | -2.0 (9.47)
  PR Interval: Change at 30 Minutes Post Last Dose | -3.0 (6.97) | -0.1 (10.26)
  QRS Duration: Change at 10 Minutes Post Last Dose | -0.8 (5.37) | -0.2 (5.35)
  QRS Duration: Change at 30 Minutes Post Last Dose | 0.9 (2.80) | -0.4 (4.05)
  QT Interval: Change at 10 Minutes Post Last Dose | -6.9 (26.28) | 0.0 (25.83)
  QT Interval: Change at 30 Minutes Post Last Dose | -8.0 (13.75) | -1.9 (23.78)
  QTcB Interval: Change at 10 Minutes Post Last Dose | 1.2 (56.80) | -3.8 (39.57)
  QTcB Interval: Change at 30 Minutes Post Last Dose | -9.3 (30.94) | -8.6 (36.21)
  QTcF Interval: Change at 10 Minutes Post Last Dose | -1.9 (44.56) | -2.5 (33.58)
  QTcF Interval: Change at 30 Minutes Post Last Dose | -8.9 (24.24) | -6.2 (30.48)
  RR Interval: Change at 10 Minutes Post Last Dose | -20.5 (138.34) | 15.9 (60.56)
  RR Interval: Change at 30 Minutes Post Last Dose | 1.6 (72.95) | 22.8 (73.59)

9. Secondary Outcome: Number of Participants by Degree of Left Ventricular Opacification (LVO) Assessed by Visual Peak Contrast Intensity
Description: LVO peak contrast intensity was determined by readers (independent blinded) using a categorical scale as None, Low, Medium, High or Blooming, where, None = Absence of contrast signal; Low = Limited capacity to make a diagnostic assessment; Presence of contrast signal does not improve diagnostic interpretability to a great degree; Medium = Good capacity to make a diagnostic assessment; Contrast signal facilitates diagnostic interpretability to a good degree; High = Optimal capacity to make a diagnostic assessment; Contrast signal facilitates diagnostic interpretability to a high degree; Blooming = Oversaturation of the signal disrupts diagnostic interpretability. Tissue boundaries become challenging to delineate. There may be excessive acoustic shadowing in the far-field of the image. Number of participants by degree of LVO assessed by visual peak contrast intensity was presented by readers and dose levels.
Time Frame: as for outcome 1
Population: PP population consisted of all participants who had available non-contrast harmonic images and OPTISON-enhanced echocardiographic images, irrespective of the quality of CE-echo and who did not have an important protocol deviation impacting study primary endpoint. Here, "Number Analyzed" signifies participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 7 | 23
Participants
  Reader 1: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 1: OPTISON Dose Level 1: None | 0 | 2
  Reader 1: OPTISON Dose Level 1: Low | 0 | 0
  Reader 1: OPTISON Dose Level 1: Medium | 2 | 8
  Reader 1: OPTISON Dose Level 1: High | 4 | 12
  Reader 1: OPTISON Dose Level 1: Blooming | 0 | 0
  Reader 1: OPTISON Dose Level 2: None | 0 | 1
  Reader 1: OPTISON Dose Level 2: Low | 0 | 0
  Reader 1: OPTISON Dose Level 2: Medium | 0 | 5
  Reader 1: OPTISON Dose Level 2: High | 7 | 16
  Reader 1: OPTISON Dose Level 2: Blooming | 0 | 1
  Reader 2: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 2: OPTISON Dose Level 1: None | 0 | 2
  Reader 2: OPTISON Dose Level 1: Low | 0 | 1
  Reader 2: OPTISON Dose Level 1: Medium | 1 | 10
  Reader 2: OPTISON Dose Level 1: High | 5 | 6
  Reader 2: OPTISON Dose Level 1: Blooming | 0 | 3
  Reader 2: OPTISON Dose Level 2: None | 0 | 1
  Reader 2: OPTISON Dose Level 2: Low | 0 | 0
  Reader 2: OPTISON Dose Level 2: Medium | 0 | 8
  Reader 2: OPTISON Dose Level 2: High | 7 | 12
  Reader 2: OPTISON Dose Level 2: Blooming | 0 | 2
  Reader 3: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 3: OPTISON Dose Level 1: None | 0 | 2
  Reader 3: OPTISON Dose Level 1: Low | 0 | 0
  Reader 3: OPTISON Dose Level 1: Medium | 3 | 9
  Reader 3: OPTISON Dose Level 1: High | 3 | 10
  Reader 3: OPTISON Dose Level 1: Blooming | 0 | 1
  Reader 3: OPTISON Dose Level 2: None | 0 | 1
  Reader 3: OPTISON Dose Level 2: Low | 0 | 1
  Reader 3: OPTISON Dose Level 2: Medium | 0 | 7
  Reader 3: OPTISON Dose Level 2: High | 7 | 14
  Reader 3: OPTISON Dose Level 2: Blooming | 0 | 0

10. Secondary Outcome: Number of Participants by Grade of Left Ventricular Opacification (LVO) Assessed by Peak Left Ventricular (LV) Contrast Filling
Description: Peak LV contrast filling for LVO was categorized as: 0 = none (0 percent [%] filling); 1 = faint (around 33% filling); 2 = intermediate (around 67% filling); 3 = full (100% filling) and data were presented by readers (independent blinded) and dose levels.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 7 | 23
Participants
  Reader 1: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 1: OPTISON Dose Level 1: None | 0 | 2
  Reader 1: OPTISON Dose Level 1: Faint | 0 | 1
  Reader 1: OPTISON Dose Level 1: Intermediate | 1 | 1
  Reader 1: OPTISON Dose Level 1: Full | 5 | 18
  Reader 1: OPTISON Dose Level 2: None | 0 | 1
  Reader 1: OPTISON Dose Level 2: Faint | 0 | 0
  Reader 1: OPTISON Dose Level 2: Intermediate | 0 | 3
  Reader 1: OPTISON Dose Level 2: Full | 7 | 19
  Reader 2: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 2: OPTISON Dose Level 1: None | 0 | 2
  Reader 2: OPTISON Dose Level 1: Faint | 0 | 0
  Reader 2: OPTISON Dose Level 1: Intermediate | 0 | 2
  Reader 2: OPTISON Dose Level 1: Full | 6 | 18
  Reader 2: OPTISON Dose Level 2: None | 0 | 1
  Reader 2: OPTISON Dose Level 2: Faint | 0 | 0
  Reader 2: OPTISON Dose Level 2: Intermediate | 0 | 2
  Reader 2: OPTISON Dose Level 2: Full | 7 | 20
  Reader 3: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 3: OPTISON Dose Level 1: None | 0 | 2
  Reader 3: OPTISON Dose Level 1: Faint | 0 | 0
  Reader 3: OPTISON Dose Level 1: Intermediate | 0 | 1
  Reader 3: OPTISON Dose Level 1: Full | 6 | 19
  Reader 3: OPTISON Dose Level 2: None | 0 | 1
  Reader 3: OPTISON Dose Level 2: Faint | 0 | 1
  Reader 3: OPTISON Dose Level 2: Intermediate | 0 | 1
  Reader 3: OPTISON Dose Level 2: Full | 7 | 20

11. Secondary Outcome: Number of Participants by Contrast Enhancement Duration in the Left Ventricular (LV) Chamber
Description: Contrast enhancement duration was determined from the time the contrast appeared in the LV to the time the contrast almost dissipated from the left chamber. 3 independent blinded reader performed evaluation.
Time Frame: as for outcome 1
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 7 | 23
Participants
  Reader 1: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 1: OPTISON Dose Level 1: 0 minute | 0 | 3
  Reader 1: OPTISON Dose Level 1: 1 minute (<1 minute contrast duration) | 1 | 2
  Reader 1: OPTISON Dose Level 1: 2 minutes (1-2 minutes contrast duration) | 3 | 5
  Reader 1: OPTISON Dose Level 1: 4 minutes (2-4 minutes contrast duration) | 2 | 10
  Reader 1: OPTISON Dose Level 1: 7 minutes (4-7 minutes contrast duration) | 0 | 2
  Reader 1: OPTISON Dose Level 1: 10 minutes (7-10 minutes contrast duration) | 0 | 0
  Reader 1: OPTISON Dose Level 1: None of the above (>10 minutes contrast duration) | 0 | 0
  Reader 1: OPTISON Dose Level 2: 0 minute | 0 | 2
  Reader 1: OPTISON Dose Level 2: 1 minute (<1 minute contrast duration) | 0 | 0
  Reader 1: OPTISON Dose Level 2: 2 minutes (1-2 minutes contrast duration) | 2 | 7
  Reader 1: OPTISON Dose Level 2: 4 minutes (2-4 minutes contrast duration) | 4 | 10
  Reader 1: OPTISON Dose Level 2: 7 minutes (4-7 minutes contrast duration) | 1 | 4
  Reader 1: OPTISON Dose Level 2: 10 minutes (7-10 minutes contrast duration) | 0 | 0
  Reader 1: OPTISON Dose Level 2: None of the above (>10 minutes contrast duration) | 0 | 0
  Reader 2: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 2: OPTISON Dose Level 1: 0 minute | 0 | 2
  Reader 2: OPTISON Dose Level 1: 1 minute (<1 minute contrast duration) | 1 | 0
  Reader 2: OPTISON Dose Level 1: 2 minutes (1-2 minutes contrast duration) | 1 | 7
  Reader 2: OPTISON Dose Level 1: 4 minutes (2-4 minutes contrast duration) | 3 | 11
  Reader 2: OPTISON Dose Level 1: 7 minutes (4-7 minutes contrast duration) | 1 | 2
  Reader 2: OPTISON Dose Level 1: 10 minutes (7-10 minutes contrast duration) | 0 | 0
  Reader 2: OPTISON Dose Level 1: None of the above (>10 minutes contrast duration) | 0 | 0
  Reader 2: OPTISON Dose Level 2: 0 minute | 0 | 1
  Reader 2: OPTISON Dose Level 2: 1 minute (<1 minute contrast duration) | 0 | 0
  Reader 2: OPTISON Dose Level 2: 2 minutes (1-2 minutes contrast duration) | 0 | 3
  Reader 2: OPTISON Dose Level 2: 4 minutes (2-4 minutes contrast duration) | 5 | 14
  Reader 2: OPTISON Dose Level 2: 7 minutes (4-7 minutes contrast duration) | 1 | 5
  Reader 2: OPTISON Dose Level 2: 10 minutes (7-10 minutes contrast duration) | 1 | 0
  Reader 2: OPTISON Dose Level 2: None of the above (>10 minutes contrast duration) | 0 | 0
  Reader 3: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 3: OPTISON Dose Level 1: 0 minute | 0 | 3
  Reader 3: OPTISON Dose Level 1: 1 minute (<1 minute contrast duration) | 2 | 2
  Reader 3: OPTISON Dose Level 1: 2 minutes (1-2 minutes contrast duration) | 1 | 7
  Reader 3: OPTISON Dose Level 1: 4 minutes (2-4 minutes contrast duration) | 3 | 10
  Reader 3: OPTISON Dose Level 1: 7 minutes (4-7 minutes contrast duration) | 0 | 0
  Reader 3: OPTISON Dose Level 1: 10 minutes (7-10 minutes contrast duration) | 0 | 0
  Reader 3: OPTISON Dose Level 1: None of the above (>10 minutes contrast duration) | 0 | 0
  Reader 3: OPTISON Dose Level 2: 0 minute | 0 | 2
  Reader 3: OPTISON Dose Level 2: 1 minute (<1 minute contrast duration) | 0 | 0
  Reader 3: OPTISON Dose Level 2: 2 minutes (1-2 minutes contrast duration) | 3 | 6
  Reader 3: OPTISON Dose Level 2: 4 minutes (2-4 minutes contrast duration) | 3 | 14
  Reader 3: OPTISON Dose Level 2: 7 minutes (4-7 minutes contrast duration) | 0 | 1
  Reader 3: OPTISON Dose Level 2: 10 minutes (7-10 minutes contrast duration) | 1 | 0
  Reader 3: OPTISON Dose Level 2: None of the above (>10 minutes contrast duration) | 0 | 0

12. Secondary Outcome: Number of Participants by Diagnostic Confidence of Left Ventricular Endocardial Border Delineation (LV EBD) and Wall Motion for Contrast and Non-Contrast Enhanced Images
Description: Diagnostic confidence for the assessment of LV EBD and wall motion was scored for non-contrast and OPTISON-enhanced echocardiographic acquisitions separately using a 4-point scale which ranged from ranged 0 to 4, where 0 = no confidence, 1 = low confidence, 2 = moderate confidence, 3 = high confidence. A higher score indicates better confidence level. Data were presented by reader (independent blinded), non-contrast and dose levels.
Time Frame: as for outcome 1
Population: PP population consisted of all participants who had available non-contrast harmonic images and OPTISON-enhanced echocardiographic images, irrespective of the quality of CE-echo and who did not have an important protocol deviation impacting study primary endpoint. Each participants underwent an echocardiographic procedure first without contrast administration, then intravenous bolus injection of OPTISON. Here, "Number Analyzed" signifies participants who were evaluable for specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 7 | 23
Participants
  Reader 1: Non-contrast: No confidence | 2 | 10
  Reader 1: Non-contrast: Low confidence | 4 | 9
  Reader 1: Non-contrast: Moderate confidence | 1 | 4
  Reader 1: Non-contrast: High confidence | 0 | 0
  Reader 1: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 1: OPTISON Dose Level 1: No confidence | 0 | 3
  Reader 1: OPTISON Dose Level 1: Low confidence | 1 | 2
  Reader 1: OPTISON Dose Level 1: Moderate confidence | 2 | 9
  Reader 1: OPTISON Dose Level 1: High confidence | 3 | 8
  Reader 1: OPTISON Dose Level 2: No confidence | 0 | 2
  Reader 1: OPTISON Dose Level 2: Low confidence | 0 | 1
  Reader 1: OPTISON Dose Level 2: Moderate confidence | 0 | 11
  Reader 1: OPTISON Dose Level 2: High confidence | 7 | 9
  Reader 2: Non-contrast: No confidence | 0 | 6
  Reader 2: Non-contrast: Low confidence | 6 | 15
  Reader 2: Non-contrast: Moderate confidence | 1 | 2
  Reader 2: Non-contrast: High confidence | 0 | 0
  Reader 2: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 2: OPTISON Dose Level 1: No confidence | 0 | 2
  Reader 2: OPTISON Dose Level 1: Low confidence | 0 | 3
  Reader 2: OPTISON Dose Level 1: Moderate confidence | 2 | 7
  Reader 2: OPTISON Dose Level 1: High confidence | 4 | 10
  Reader 2: OPTISON Dose Level 2: No confidence | 0 | 2
  Reader 2: OPTISON Dose Level 2: Low confidence | 0 | 1
  Reader 2: OPTISON Dose Level 2: Moderate confidence | 1 | 10
  Reader 2: OPTISON Dose Level 2: High confidence | 6 | 10
  Reader 3: Non-contrast: No confidence | 1 | 10
  Reader 3: Non-contrast: Low confidence | 2 | 7
  Reader 3: Non-contrast: Moderate confidence | 3 | 5
  Reader 3: Non-contrast: High confidence | 1 | 1
  Reader 3: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 3: OPTISON Dose Level 1: No confidence | 0 | 2
  Reader 3: OPTISON Dose Level 1: Low confidence | 0 | 2
  Reader 3: OPTISON Dose Level 1: Moderate confidence | 3 | 7
  Reader 3: OPTISON Dose Level 1: High confidence | 3 | 11
  Reader 3: OPTISON Dose Level 2: No confidence | 0 | 1
  Reader 3: OPTISON Dose Level 2: Low confidence | 0 | 0
  Reader 3: OPTISON Dose Level 2: Moderate confidence | 2 | 11
  Reader 3: OPTISON Dose Level 2: High confidence | 5 | 11

13. Secondary Outcome: Number of Participants by Diagnostic Confidence of Left Ventricular Ejection Fraction (LVEF) for Non-contrast and OPTISON Enhanced Echocardiography
Description: Diagnostic confidence for the evaluation of LVEF was calculated using the formula: (end diastole volume - end systole volume)/(end diastole volume) was scored for non-contrast and OPTISON-enhanced echocardiographic acquisitions separately using a 4-point scale which ranged from 0 to 3, where 0 = no confidence, 1 = low confidence, 2 = moderate confidence, 3 = high confidence. A higher score indicates better confidence level. Data were presented by reader (independent blinded), non-contrast and dose levels.
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
Number analyzed (Participants) | 7 | 23
Participants
  Reader 1: Non-contrast: No confidence | 4 | 11
  Reader 1: Non-contrast: Low confidence | 3 | 11
  Reader 1: Non-contrast: Moderate confidence | 0 | 1
  Reader 1: Non-contrast: High confidence | 0 | 0
  Reader 1: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 1: OPTISON Dose Level 1: No confidence | 0 | 5
  Reader 1: OPTISON Dose Level 1: Low confidence | 1 | 1
  Reader 1: OPTISON Dose Level 1: Moderate confidence | 2 | 10
  Reader 1: OPTISON Dose Level 1: High confidence | 3 | 6
  Reader 1: OPTISON Dose Level 2: No confidence | 0 | 2
  Reader 1: OPTISON Dose Level 2: Low confidence | 0 | 1
  Reader 1: OPTISON Dose Level 2: Moderate confidence | 0 | 11
  Reader 1: OPTISON Dose Level 2: High confidence | 7 | 9
  Reader 2: Non-contrast: No confidence | 2 | 16
  Reader 2: Non-contrast: Low confidence | 3 | 5
  Reader 2: Non-contrast: Moderate confidence | 2 | 2
  Reader 2: Non-contrast: High confidence | 0 | 0
  Reader 2: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 2: OPTISON Dose Level 1: No confidence | 0 | 4
  Reader 2: OPTISON Dose Level 1: Low confidence | 0 | 0
  Reader 2: OPTISON Dose Level 1: Moderate confidence | 2 | 10
  Reader 2: OPTISON Dose Level 1: High confidence | 4 | 8
  Reader 2: OPTISON Dose Level 2: No confidence | 0 | 2
  Reader 2: OPTISON Dose Level 2: Low confidence | 0 | 1
  Reader 2: OPTISON Dose Level 2: Moderate confidence | 1 | 8
  Reader 2: OPTISON Dose Level 2: High confidence | 6 | 12
  Reader 3: Non-contrast: No confidence | 3 | 17
  Reader 3: Non-contrast: Low confidence | 0 | 3
  Reader 3: Non-contrast: Moderate confidence | 2 | 3
  Reader 3: Non-contrast: High confidence | 2 | 0
  Reader 3: OPTISON Dose Level 1: number analyzed (Participants) | 6 | 22
  Reader 3: OPTISON Dose Level 1: No confidence | 0 | 4
  Reader 3: OPTISON Dose Level 1: Low confidence | 2 | 5
  Reader 3: OPTISON Dose Level 1: Moderate confidence | 1 | 7
  Reader 3: OPTISON Dose Level 1: High confidence | 3 | 6
  Reader 3: OPTISON Dose Level 2: No confidence | 1 | 7
  Reader 3: OPTISON Dose Level 2: Low confidence | 0 | 1
  Reader 3: OPTISON Dose Level 2: Moderate confidence | 1 | 6
  Reader 3: OPTISON Dose Level 2: High confidence | 5 | 9

ADVERSE EVENTS:
Time Frame: 0- 72 hours
Description: The Safety population consisted of all enrolled participants who received >=1 dose of OPTISON in the study.
Groups:
- Body Weight Group <=40 kg: OPTISON: Participants with body weight >=20 to <=28 kg received OPTISON 0.1 mL (dose level 1) or 0.2 mL (dose level 2); and participants with body weight >28 to <=40 kg received OPTISON 0.2 mL (dose level 1) or 0.3 mL (dose level 2) IV injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose for body weight >=20 to <=28 kg and >28 to <=40 kg was 1.0 mL and 1.5 mL per dose level, respectively.
  All subjects were imaged without contrast then with dose level 1 and then dose level 2. So it is impossible to separate the AE for each intervention.
- Body Weight Group >40 kg: OPTISON: Participants with body weight >40 kg received OPTISON 0.2 (dose level 1) or 0.4 mL (dose level 2) IV injection, 10 minutes apart on Day 1. The maximum allowed cumulative dose was 1.8 mL per dose level.
  All subjects were imaged without contrast then with dose level 1 and then dose level 2. So it is impossible to separate the AE for each intervention.
Arm/Group | Body Weight Group <=40 kg: OPTISON | Body Weight Group >40 kg: OPTISON
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/29
Other Adverse Events (participants affected / at risk) | 4/8 | 9/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Body Weight Group <=40 kg: OPTISON (N=8) | Body Weight Group >40 kg: OPTISON (N=29)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 3
Migraine (Nervous system disorders) | 0 | 1
Taste disorder (Nervous system disorders) | 1 | 1
Mood swings (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI and/or institution is that the Sponsor can review results communications prior to public release and can restrict communications regarding trial results for a period that is more than 30 days (publications/abstracts) but not to exceed 90 days (patent related issues) from the time submitted to the Sponsor to review. The PI may be asked to remove any Sponsor confidential information and/or delay publication to protect any proprietary information.

DOCUMENTS (2):
  • Study Protocol (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT03740997/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT03740997/SAP_001.pdf